CLINICAL TRIAL: NCT05741606
Title: Evaluation of the Safety and Efficacy and of Sodium Pentaborate Pentahydrate in People With Overweight and Obesity: a Randomized, Double-blind, Placebo-controlled Phase 1/2 Trial
Brief Title: Safety and Efficacy of Sodium Pentaborate Pentahydrate in People With Overweight and Obesity
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Saeid Safiri, Principal Investigator, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 70928
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Sodium pentaborate pentahydrate
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Capsules containing sodium pentaborate pentahydrate 200 mg (Active Comparator): Capsules containing sodium pentaborate pentahydrate 200 mg orally once a day
  Interventions: Drug: Sodium pentaborate pentahydrate
- Capsules containing sodium pentaborate pentahydrate 400 mg (Active Comparator): Capsules containing sodium pentaborate pentahydrate 400 mg orally once a day
  Interventions: Drug: Sodium pentaborate pentahydrate
- Capsules containing sodium pentaborate pentahydrate 600 mg (Active Comparator): Capsules containing sodium pentaborate pentahydrate 600 mg orally once a day
  Interventions: Drug: Sodium pentaborate pentahydrate
- Capsules containing sodium pentaborate pentahydrate 800 mg (Active Comparator): Capsules containing sodium pentaborate pentahydrate 800 mg orally once a day
  Interventions: Drug: Sodium pentaborate pentahydrate
- Capsules containing sodium pentaborate pentahydrate 1000 mg (Active Comparator): Capsules containing sodium pentaborate pentahydrate 1000 mg orally once a day
  Interventions: Drug: Sodium pentaborate pentahydrate
- Placebo capsules (Placebo Comparator): Placebo capsules of the same shape, smell, and color orally once a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium pentaborate pentahydrate — Capsules containing sodium pentaborate pentahydrate 200, 400, 600, 800, and 1000 mg
  Arms: Capsules containing sodium pentaborate pentahydrate 1000 mg; Capsules containing sodium pentaborate pentahydrate 200 mg; Capsules containing sodium pentaborate pentahydrate 400 mg; Capsules containing sodium pentaborate pentahydrate 600 mg; Capsules containing sodium pentaborate pentahydrate 800 mg
Drug: Placebo — Placebo capsules
  Other Names: Placebo capsules
  Arms: Placebo capsules

SUMMARY:
This study investigates the safety and efficacy of sodium pentaborate pentahydrate in improving the body weight and glycemic profile of patients with overweight or obesity compared to the placebo group.

DETAILED DESCRIPTION:
Obesity is considered one of the pandemics of the current century which is associated with great mortality and morbidity. In addition to changing diet and physical activity, medicines, devices, and even surgery are suggested for obesity. Although they can be effective partially, however, the rate of recurrence is high and some are invasive. So, there is a need to evaluate other types of potential interventions for obesity management. Due to the effects of boron-derivates in the prevention and management of obesity, we will evaluate the safety and efficacy of sodium pentaborate pentahydrate in patients with overweight and obesity in terms of its safety and efficacy. This study will be conducted as a randomized, double-blind, placebo-controlled, parallel-group, dose-ranging, phase 1/2 trial. Individuals aged ≥18 years with body mass index (BMI) ≥30.0 kg/m2 or BMI ≥27.0 kg/m2 with the presence of hypertension or dyslipidemia will be recruited. Participants will be randomly assigned (6:1) to oral administration of once-daily sodium pentaborate pentahydrate (200, 400, 600, 800, 1000 mg), or placebo, using balanced block randomization. The primary endpoint will be the relative change from baseline in body weight (%) at 12 weeks. Adverse events will be monitored and checked closely in terms of physical examinations and laboratory measures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing the informed consent.
* A non-pregnant female participant or a male participant who has been surgically sterilized (vasectomy) or is willing to use appropriate contraceptive methods during the trial (until the end of the trial).
* Body mass index (BMI) ≥30·0 kg/m2 or BMI ≥27·0 kg/m2 in the presence of hypertension or dyslipidemia (treated or untreated, assessed at the discretion of the investigator).

Exclusion Criteria:

* Glycosylated hemoglobin (HbA1c) ≥48 mmol/mol (6.5%) as measured by the laboratory at screening.
* History of type 1 or type 2 diabetes.
* Treatment with glucose-lowering drug(s) within 90 days prior to screening.
* Obesity caused by endocrine disorders (such as Cushing's syndrome)
* Change in body weight of more than 5 kg during the 90 days before screening regardless of medical records.
* Treatment with any drug proven to control weight in the 90 days before screening.
* Previous or planned obesity treatment (during the trial period) with surgery or a weight loss device. However, the following are permitted: (1) liposuction and/or abdominoplasty, if performed more than one year prior to screening; (2) lap banding, if the banding was removed more than 1 year before the screening. (3) intragastric balloon, if the balloon was removed more than 1 year before the screening. or (4) duodenal-jejunal bypass sleeve, if the sleeve was removed more than 1 year before the screening.
* Uncontrolled thyroid disease, defined as TSH >4·78 mIU/L or 1.5 times the upper limit of normal as measured by a laboratory at screening.
* Inadequately treated hypertension, defined at screening as systolic ≥180 mmHg or diastolic ≥110 mmHg.
* History of malignant neoplasms in the last 5 years before the screening. Basal and squamous cell skin cancer and any in situ cancer are allowed.
* Presence or history of cardiovascular disease, including stable and unstable angina pectoris, myocardial infarction, transient ischemic attack, stroke, cardiac decompensation, clinically significant arrhythmias, or clinically significant conduction disturbances.
* The participant is currently classified as having New York Heart Association Class IV heart failure.
* Surgery planned during the trial period, excluding minor surgery, at the discretion of the investigator.
* Known or suspected abuse of alcohol or recreational drugs.
* Known or suspected hypersensitivity to test product(s) or related products.
* Participation in another clinical trial within 90 days prior to screening.
* Personal or first-degree relative history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.
* Presence of acute pancreatitis within 180 days before screening.
* History or presence of chronic pancreatitis.
* Any impairment, unwillingness, or disability, not covered by any of the other exclusion criteria, that in the opinion of the investigator may compromise the participant's safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-21 (Estimated); Primary Completion 2024-03-20 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
Change of body weight | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  The relative change of body weight compared to the base weight (%)

SECONDARY OUTCOMES:
Weight loss ≥ 5% of initial body weight | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Proportion (%) of people with weight loss ≥ 5% of initial body weight
Weight loss ≥ 10% of initial body weight | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Proportion (%) of people with weight loss ≥ 10% of initial body weight
Change in waist circumference | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Relative change in waist circumference compared to baseline
Change in body mass index | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Relative change in body mass index compared to baseline
Change of waist to hip circumference | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Relative change of waist to hip circumference compared to baseline
Hemoglobin A1c level | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Change in hemoglobin A1c level
Fasting blood glucose | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Change in fasting blood glucose levels
Insulin level | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Change in insulin level
Systolic and diastolic blood pressures | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Changes in systolic and diastolic blood pressures
High density lipoprotein (HDL) levels | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Changes in high density lipoprotein (HDL) levels
Low density lipoprotein (LDL) levels | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Changes in low density lipoprotein (LDL) levels
Triglyceride levels | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Changes in triglyceride levels
Total cholesterol levels | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Changes in total cholesterol levels
High-sensitivity C-reactive protein levels | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Changes in high-sensitivity C-reactive protein levels
Short-Form 36 (SF-36) v2·0 acute score | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Changes in Short-Form 36 (SF-36) v2·0 acute scores. It ranges zero to 100 and lower scores mean higher disability.
Three-Factor Eating Questionnaire Revised 18-item version 2 score (TFEQ-R18v2) | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Changes in Three-Factor Eating Questionnaire Revised 18-item version 2 score (TFEQ-R18v2). It has four-point response scales ranging from definitely true (score = 4) to definitely false (score = 1).
Adverse events | Screening, randomization and weeks 2, 4, 6, 8, 10, 12, 16
  Registration of adverse events in questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Saeid Safiri, PhD, Principal Investigator — Tabriz University of Medical Sciences
Locations (1):
- Imam Reza hospital and Clinic of Salamat, Tabriz, East Azarbayejan, Iran

IPD SHARING:
Plan to Share IPD: No